CLINICAL TRIAL: NCT00642746
Title: Phase II Study of Erlotinib (Tarceva) Alternating With Chemotherapy for Second-line Treatment of Metastatic Colorectal Cancer With Molecular Correlates for p53 Pathway
Brief Title: Erlotinib and Chemotherapy for 2nd Line Treatment (Tx) of Metastatic Colorectal Cancer (mCRC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor enrollment and grade 3 toxicities noted during an interim analysis.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3753
Record Dates: First submitted 2008-03-24; First posted 2008-03-25 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colon; Cancer; Metastatic; Colorectal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Erlotinib Hydrochloride; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX with Erlotinib (Experimental): Subjects received FOLFOX (Leucovorin, Fluorouracil, and Oxaliplatin) and Erlotinib. Treatment consisted of a 28 day cycle. Subjects received FOLFOX on days 1, 2, and 3, and 15-16, followed by Erlotinib on days 3-8, and 17-22.
  Interventions: Drug: Erlotinib; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- FOLFIRI with Erlotinib (Experimental): Subjects received FOLFIRI (Leucovorin, Fluorouracil, and Irinotecan) and Erlotinib. Treatment consisted of a 28 day cycle. Subjects received FOLFIRI on days 1, 2, and 3, and 15-16, followed by Erlotinib on days 3-8, and 17-22.
  Interventions: Drug: Erlotinib; Drug: Fluorouracil; Drug: Leucovorin; Drug: Irinotecan

INTERVENTIONS:
Drug: Erlotinib — Erlotinib oral tablets are conventional, immediate-release tablets containing erlotinib as the hydrochloride salt. In addition to the active ingredient, erlotinib contains lactose (hydrous), microcrystalline cellulose, sodium starch glycolate, sodium lauryl sulfate, and magnesium stearate.
  Tablets containing 25 mg, 100 mg, and 150 mg of erlotinib are available. Each bottle will contain 30 tablets, a quantity sufficient for 4 consecutive weeks of dosing, with overage.
  Other Names: Tarceva
Drug: Fluorouracil — Antimetabolite used as a chemotherapy. Administered intravenously as a bolus injection at 400mg/m2 on Day 1 followed by 2400 mg/m2 continuously over 46 hours.
Drug: Leucovorin — Chemotherapy agent given as a supplement to Fluorouracil. Given intravenously 400mg/m2 in combination with Fluorouracil dosing.
Drug: Oxaliplatin — Platinum-based antineoplastic chemotherapy agent given intravenously at 85 mg/m2.
  Arms: FOLFOX with Erlotinib
Drug: Irinotecan — Chemotherapy agent given intravenously at 180 mg/m2.
  Arms: FOLFIRI with Erlotinib

SUMMARY:
The purpose of this study is to see if alternating chemotherapy with erlotinib increases tumor shrinkage in people with metastatic colorectal cancer. The investigator will also be studying the side effects (good and bad) of alternating chemotherapy with erlotinib on metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria to be eligible for study entry:

* Age 18-80
* Able to provide informed consent
* Biopsy proven unresectable metastatic adenocarcinoma of the colon or rectum
* Documented progression on prior first-line oxaliplatin-based or irinotecan-based regimen for metastatic colorectal cancer
* Radiographically measurable disease with at least one bidimensionally measurable lesion of > 1 cm
* Prior first-line regimen must have been completed at least 4 weeks prior to study treatment
* Use of biologic agents with first-line chemotherapy permitted
* Previous adjuvant regimens must have been greater than 6 months before inclusion
* Adequate organ function including bone marrow, liver and renal function as defined by the following values: absolute neutrophil count > 1500/microliter; Hgb > 9 g/dL; platelets > 90,000/microliter; International Normalized Ratio < 1.8 (unless in therapeutic range if taking warfarin or other warfarin-derivative anticoagulants and are being monitored regularly for changes in prothrombin time or International Normalized Ratio); bilirubin < 2 times the Upper Limit of Normal; alkaline phosphatase < 3 times the Upper Limit of Normal; aspartate aminotransferase/alanine aminotransferase < 5 times the Upper Limit of Normal; serum creatinine < 1.5 times the Upper Limit of Normal
* Eastern Cooperative Oncology Group status < 2

Exclusion Criteria:

Patients meeting any of the following criteria are ineligible for study entry:

* Prior second-line chemotherapy regimens for colorectal cancer
* Prior treatment with erlotinib or gefitinib
* Central Nervous System metastasis
* Second malignancies less than 5 years prior to enrollment. Completely resected basal or squamous cell carcinoma of the skin is allowed.
* Untreated/unresolved bowel obstruction
* Inability to take oral mediations
* HIV positive
* Pregnancy
* Other uncontrolled medical illnesses
* Current diarrhea > grade 2
* Symptomatic angina or uncontrolled congestive heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was done from 3/28/2008 to the study closure of 12/19/2011. Patients were recruited from the Oregon Health and Science University medical clinic as well as via referral from associated regional medical clinics.
Pre-assignment Details: Patients were stratified according to whether they had received 5-Fluorouracil/Leucovorin with Oxaliplatin or Fluorouracil, Leucovorin, and Irinotecan for their 1st line treatment. Whichever they had not received in the 1st line setting, they received on trial. 16 patients signed consent. 2 patients withdrew, 3 ineligible, and 1 unevaluable.
Period: Overall Study
Arm/Group | FOLFIRI With Erlotinib | FOLFOX With Erlotinib
Started | 10 | 1
Completed | 9 | 1
Not Completed | 1 | 0
Not completed — Patient unevaluable | 1 | 0

BASELINE CHARACTERISTICS:
Population: 11 patients included for all baseline measures except for age, categorical because the age is missing for the 1 patient who eventually was ineligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFIRI With Erlotinib | FOLFOX With Erlotinib | Total
Number analyzed (Participants) | 10 | 1 | 11
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 7
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Response Rates of Radiographically Measurable Disease
Description: The primary outcome measure will be the response rates of radiographically measurable disease. Response rate of disease will be assessed per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), >= 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: Disease response assessed after every 2 Treatment Cycles, or around 8 weeks.
Population: Patients who were considered for analysis were those who received treatment in a manner consistent with the protocol, as determined by the investigator.
Measure: Number; unit: Number of Patients
Arm/Group | FOLFIRI With Erlotinib | FOLFOX With Erlotinib
Number analyzed (Participants) | 10 | 1
Number of Patients
  Best Outcome - Complete Response | 0 | 0
  Best Outcome - Partial Response | 1 | 0
  Best Outcome- Stable Disease | 5 | 1
  Best Outcome - Progressive Disease | 4 | 0

2. Secondary Outcome: Second-line Progression Free Survival
Description: Time to disease progression from start of second-line experimental regimen. Disease progression will be measured per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), >= 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: Upon completion of follow-up, for an average of 99 days following the initiation of study treatment.
Population: Patients who were considered for analysis were those who received treatment in a manner consistent with the protocol, as determined by the investigator.
  95% CI cannot be computed for FOLFOX with Erlotinib arm because there is only one patient.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | FOLFIRI With Erlotinib | FOLFOX With Erlotinib
Number analyzed (Participants) | 10 | 1
Days | 83 [15 to 127] | 125

3. Secondary Outcome: Time to Second Progression (From Start of First-Line Regimen)
Description: Number of days from the initiation of first line treatment to first documented progression. Progression will be assessed per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), >= 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
  Progression free survival (time to progression or death, whichever occurs first) is the same as time to progression as all of the patients in this trial progressed.
Time Frame: Documented by Follow-up CT scans following first line treatment, average of 225 days.
Population: 95% CI cannot be computed for FOLFOX with Erlotinib arm because there is only one patient.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | FOLFIRI With Erlotinib | FOLFOX With Erlotinib
Number analyzed (Participants) | 10 | 1
Days | 83 [15 to 127] | 125

ADVERSE EVENTS:
Time Frame: Adverse Events have been collected since the study opened to enrollment to study closure, totaling 5.5 years.
Arm/Group | FOLFIRI With Erlotinib | FOLFOX With Erlotinib
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/1
Other Adverse Events (participants affected / at risk) | 8/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRI With Erlotinib (N=9) | FOLFOX With Erlotinib (N=1)
GI Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 — Patient admitted with GI hemorrhage and malignant ascites, attributed to his underlying disease.
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 — Patient admitted with GI hemorrhage and malignant ascites, attributed to his underlying disease.
Weakness (General disorders) | 1 (1) | 0 (0) — Patient admitted for weakness, fatigue, leukopenia, hyperbilirubinemia, and thrombocytopenia. All related to Fluorouracil, Leucovorin, and Irinotecan , and possibly related to Erlotinib, per the Investigator.
Fatigue (General disorders) | 1 (1) | 0 (0) — Patient admitted for weakness, fatigue, leukopenia, hyperbilirubinemia, and thrombocytopenia. All related to Fluorouracil, Leucovorin, and Irinotecan , and possibly related to Erlotinib, per the Investigator.
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Patient admitted for weakness, fatigue, leukopenia, hyperbilirubinemia, and thrombocytopenia. All related to Fluorouracil, Leucovorin, and Irinotecan, and possibly related to Erlotinib, per the Investigator.
Hyperbilirubinemia (Investigations) | 1 (1) | 0 (0) — Patient admitted for weakness, fatigue, leukopenia, hyperbilirubinemia, and thrombocytopenia. All related to Fluorouracil, Leucovorin, and Irinotecan, and possibly related to Erlotinib, per the Investigator.
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Patient admitted for weakness, fatigue, leukopenia, hyperbilirubinemia, and thrombocytopenia. All related to Fluorouracil, Leucovorin, and Irinotecan, and possibly related to Erlotinib, per the Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRI With Erlotinib (N=9) | FOLFOX With Erlotinib (N=1)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) — Grade 3 or 4 Neutropenia while on trial.
Oral Pain (General disorders) | 2 (2) | 0 (0) — Grade 3 or 4 Oral Pain
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Diarrhea
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Nausea
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Rash
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Hyponatremia
International Normalized Ratio Elevation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 3 or 4
Abdominal Pain (General disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Abdominal Pain
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3 or 4 GI Bleed
Fatigue (General disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Fatigue
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Leukopenia

LIMITATIONS AND CAVEATS:
Study terminated before target enrollment was reached due to excessive toxicities and limited enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes